CLINICAL TRIAL: NCT07229066
Title: Evaluation of the Effect of Video-Based Education on Bowel Preparation Before Colonoscopy
Brief Title: The Effect of Video-Based Education on Colonoscopy Preparation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Şafak Meric Ozgenel, Assistant Professor Dr., Eskisehir Osmangazi University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: ESOGU-OZGENEL-2025-COLONOSCOPY
Record Dates: First submitted 2025-11-13; First posted 2025-11-14 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Bowel Preparation Quality; Colonoscopy; Patient Education

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to either a video-based education group or a control group receiving standard written and verbal instructions. Both groups will be followed in parallel to assess the effect of the intervention on bowel preparation quality before colonoscopy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Video-based education group for Sodium Picosulfate (0.1 g) sennoside b (3 mg) + Bisacodyl (5 mg) (Experimental): Participants receive a video-based education program explaining colonoscopy preparation steps, diet instructions, and use of laxatives.
  Interventions: Behavioral: Video Education
- Control group for Sodium Picosulfate (0.1 g) sennoside B (3 mg) + Bisacodyl (5 mg) (No Intervention): Participants receive routine written and verbal instructions for colonoscopy preparation.
- Video-based education group for Sodium Picosulfate (0.1 g) (Experimental): Participants receive a video-based education program explaining colonoscopy preparation steps, diet instructions, and use of laxatives.
  Interventions: Behavioral: Video Education
- Control group for Sodium Picosulfate (0.1 g) (No Intervention): Participants receive routine written and verbal instructions for colonoscopy preparation.
- Video-based education group for Sennoside A+B (1875 mg) (Experimental): Participants receive a video-based education program explaining colonoscopy preparation steps, diet instructions, and use of laxatives.
  Interventions: Behavioral: Video Education
- Control group for Sennoside A+B (1875 mg) (No Intervention): Participants receive routine written and verbal instructions for colonoscopy preparation.

INTERVENTIONS:
Behavioral: Video Education — Participants receive routine written and verbal instructions about colonoscopy preparation, including dietary instructions and use of prescribed laxatives. This represents the standard care provided at the study site.
  Arms: Video-based education group for Sennoside A+B (1875 mg); Video-based education group for Sodium Picosulfate (0.1 g); Video-based education group for Sodium Picosulfate (0.1 g) sennoside b (3 mg) + Bisacodyl (5 mg)

SUMMARY:
Colonoscopy is a routine procedure for evaluating gastrointestinal symptoms, detecting colorectal cancer, and removing polyps. Its effectiveness depends on patient compliance with bowel preparation instructions. However, inadequate bowel preparation occurs in 20-25% of colonoscopies, often due to non-adherence, medical conditions, or long waiting times. Poor preparation can reduce examination quality, prevent detection of precancerous lesions, and increase healthcare costs. Video-based education has been shown to be more effective than written or verbal instructions in improving bowel preparation. This study aims to evaluate the effect of video-based education on colonoscopy bowel preparation and contribute evidence to optimize patient compliance.

DETAILED DESCRIPTION:
Colonoscopy is a standard procedure performed for the evaluation of gastrointestinal symptoms, colorectal cancer screening, polyp detection, and polyp removal. Colorectal cancer (CRC) is the second leading cause of cancer-related deaths in the United States , and in Türkiye, 21,718 new cases were reported in 2022. These statistics underscore the importance of colonoscopy as a preventive and diagnostic tool.

When conducted properly, colonoscopy is safe and well-tolerated, allowing visualization of the entire colon and distal terminal ileum. The procedure's optimal effectiveness relies heavily on patient compliance with bowel preparation instructions. Unfortunately, inadequate bowel preparation occurs in approximately 20-25% of colonoscopies, often due to non-adherence, medical conditions affecting bowel cleansing, or prolonged waiting times for the procedure.

While interventions addressing medical conditions or waiting times may not always be feasible, non-compliance with preparation instructions represents a modifiable, patient-related factor. Effective bowel preparation requires adherence to dietary recommendations and the use of prescribed laxatives. The quality of preparation impacts examination adequacy, procedure duration, cancellation rates, and the need for repeat colonoscopies. Inadequate preparation can hinder thorough evaluation, prevent detection of precancerous lesions such as polyps, and increase healthcare costs.

Emerging evidence suggests that video-based educational interventions are more effective than traditional written or verbal instructions, phone calls, social media applications, or messaging services in improving patient compliance and bowel preparation quality.

This study aims to assess the effect of video-based education on bowel preparation before colonoscopy. By evaluating its impact on preparation quality and patient adherence, the study seeks to provide evidence for implementing more effective educational strategies in colonoscopy units, thereby optimizing clinical outcomes and resource utilization.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary participation in the study.
* Outpatient follow-up.
* No prior history of colonoscopy.
* Participant or a household member (spouse, child, parent, sibling) owns and can use a smartphone application.

Exclusion Criteria:

* History of major abdominal surgery.
* Suspected obstructive lesion in the gastrointestinal tract on cross-sectional imaging.
* Impaired swallowing reflex.
* Mental disorder.
* Communication difficulties (speech, perception, comprehension problems).
* Congestive heart failure or kidney failure.
* Pregnancy or breastfeeding.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Quality of Bowel Preparation | Day of Colonoscopy
  The quality of bowel preparation will be assessed on the day of colonoscopy using the Boston Bowel Preparation Scale (BBPS). This scale evaluates cleansing in three segments of the colon. Higher scores indicate better preparation, reflecting patient compliance with dietary and laxative instructions and the effectiveness of the educational intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Eskisehir Osmangazi University, Eskişehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
All requested data can be shared.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: End date of the study and one year after that
Access Criteria: The paper reviewers will be able to access the IPD and supporting information.

REFERENCES:
- [Result] Walker TB, Hengehold TA, Garza K, Rogers BD, Early D. An Interactive Video Educational Tool Does Not Improve the Quality of Bowel Preparation for Colonoscopy: A Randomized Controlled Study. Dig Dis Sci. 2022 Jun;67(6):2347-2357. doi: 10.1007/s10620-021-07215-8. Epub 2021 Aug 25. PMID 34435269
- [Result] Chan WK, Saravanan A, Manikam J, Goh KL, Mahadeva S. Appointment waiting times and education level influence the quality of bowel preparation in adult patients undergoing colonoscopy. BMC Gastroenterol. 2011 Jul 28;11:86. doi: 10.1186/1471-230X-11-86. PMID 21798022